CLINICAL TRIAL: NCT01501968
Title: Efficacy of Ascorbic Acid for Prevention of Colistin-Associated Nephrotoxicity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEU 2012-01
Record Dates: First submitted 2011-12-24; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Drug Safety
Keywords: Colistin; ascorbic acid; renal toxicity
MeSH Terms: interventions — Colistin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colistin (Active Comparator): Colistimethate sodium 2.5-5mg/kg iv
  Interventions: Drug: Colistin
- Colistin + Ascorbic acid (Experimental): Colistimethate sodium 2.5-5mg/kg iv and ascorbic acid 2 grams iv every 12 hours
  Interventions: Drug: Colistin + Ascorbic acid

INTERVENTIONS:
Drug: Colistin — Colistimethate sodium 2.5-5mg/kg iv per day
  Other Names: Colistate
  Arms: Colistin
Drug: Colistin + Ascorbic acid — Colistimethate sodium 2.5-5mg/kg iv per day and ascorbic acid 2 grams iv q 12 hours
  Other Names: vitamin c
  Arms: Colistin + Ascorbic acid

SUMMARY:
Ascorbic acid (Vitamin C) could protect renal toxicity from colistin.

DETAILED DESCRIPTION:
Renal toxicity due to colistin therapy is common. Ascorbic acid (vitamin C) has been shown to prevent colistin associated renal toxicity in animals. This study is conducted to determine if acorbic acid can prevent Colistin-Associated Nephrotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years hospitalized patient who needs colistin for therapy of nosocomial infection

Exclusion Criteria:

* pregnant woman
* lactating mother
* allergy to ascorbic acid
* receiving non-steroidal antiinflammatory drugs (NSAID), aminoglycosides, vancomycin, cisplatin, amphotericin-B
* received radiocontrast media within 1 week
* renal stone
* G-6-PD deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with Renal toxicity associated with colistin | up to 28 days
  Renal toxicity associated with colistin according to RIFLE criteria

SECONDARY OUTCOMES:
number of subjects with cure or improvement | up to 28 days
  cure improvement worse death

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Sirijatuphat R, Limmahakhun S, Sirivatanauksorn V, Nation RL, Li J, Thamlikitkul V. Preliminary clinical study of the effect of ascorbic acid on colistin-associated nephrotoxicity. Antimicrob Agents Chemother. 2015;59(6):3224-32. doi: 10.1128/AAC.00280-15. Epub 2015 Mar 23. PMID 25801556
- See also: mahidol webpage — http://mahidol.ac.th